CLINICAL TRIAL: NCT01610934
Title: Phase 2 Study: A Double-blind, Randomised, Clinical Cross-over Trial to Investigate the Treatment Potential of Liraglutide Compared to Glimepiride in MODY Patients
Brief Title: The Effects of GLP-1 in Maturity-Onset Diabetes of The Young (MODY)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: Novo Nordisk A/S (Industry); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Signe H Østoft, MD, MD, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MODY-TREAT; 2012-000592-17 (EudraCT Number)
Record Dates: First submitted 2012-05-24; First posted 2012-06-04 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Maturity-onset Diabetes of the Young
Keywords: MODY; Monogenic diabetes; Non-autoimmune diabetes; MODY3
MeSH Terms: conditions — Mason-Type Diabetes; Diabetes Mellitus, Type 2; Maturity-Onset Diabetes of the Young, Type 3 | interventions — Liraglutide; glimepiride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- liraglutide (Experimental)
  Interventions: Drug: liraglutide
- glimepiride (Active Comparator)
  Interventions: Drug: Glimepiride

INTERVENTIONS:
Drug: liraglutide — The initial daily dose will be 0.6 mg for one week, 1.2 mg the following week and then 1.8 mg for the remaining treatment period. Patients who, due to adverse events, do not tolerate up-titration to 1.8 mg liraglutide will remain on 1.2 mg of liraglutide. The injection is administered once daily in the morning.
  Other Names: Victoza®
  Arms: liraglutide
Drug: Glimepiride — At randomisation patients will be initiated on their pre-study daily dose of glimepiride minus 0.5 mg. After one week the dose will be titrated (see below). Drug naïve patients will be initiated on an initial dosage of glimepiride of 0.5 mg for one week. Thereafter, glimepiride is increased to 1.0 mg and after another one week to 1.5 mg, and there after further up to 3 mg (if the average FPG during one week is above 6 mM). The dose of glimepiride can be increased up to 4 mg if average FPG is above 6 mM and no symptoms of hypoglycaemia are observed.
  Other Names: Amaryl®
  Arms: glimepiride

SUMMARY:
The purpose of this study is to evaluate the treatment potential of GLP-1-analogues in patients with Maturity Onset Diabetes of the Young (MODY) compared to common treatment.

DETAILED DESCRIPTION:
Maturity-onset diabetes of the young (MODY) is a monogenic form of diabetes responsible for approximately 1-2% of all cases of diabetes. The disease is clinically defined by: 1) autosomal dominant inheritance (diabetes for at least two consecutive generations), 2) non-insulin dependent diabetes at onset (or measurable serum C-peptide three years after onset), and 3) diagnosis in a young age (at least one family member with onset before the age of 25 years). Clinically, MODY-patients resemble patients with type 2 diabetes (T2DM) more than patients with type 1 diabetes mellitus (T1DM). MODY is genetically heterogeneous, with known mutations in eight different genes and mutations in either of these genes leads to specific forms of MODY. Based on a national epidemiological survey, we know that in Denmark, approximately 50% of patients who are diagnosed with MODY have mutations in the hepatocyte nuclear factor (HNF) 4 alpha (HNF4A) (MODY1), glucokinase (GCK) (MODY2), or HNF1A (MODY3) genes.

MODY3 is the most common form of MODY in Denmark (approximately 60% of all patients with MODY). Patients with MODY3 are often diagnosed around puberty, more than 50% of mutation carriers will develop diabetes before the age of 25, and the lifetime risk of developing diabetes is higher than 95%. The typical course of disease is characterised by a rapid progression from impaired glucose tolerance to diabetes. After the diagnosis of diabetes, the glucose tolerance is further impaired due to a continuous loss of beta cell function. MODY3 often develops abruptly with classic hyperglycaemic symptoms such as polyuria and polydipsia, which is why this form of diabetes is often misclassified as T1DM. Patients with MODY3 have the same risk of developing microvascular and macrovascular late diabetic complications as patients with T2DM, and, strict glycaemic control combined with proper screening for diabetic late complications is crucial for a good prognosis.

About half of MODY3 patients are treated with diet or oral antidiabetic agents, the latter mostly in the form of sulphonylureas (SU), which, if possible is preferred to insulin injections. Due to a high sensitivity to SU combined with normal or even increased insulin sensitivity (MODY3 patients are more insulin sensitive than age- and body mass index (BMI)-matched patients with T2DM), this treatment is often associated with hypoglycaemia even when rather low doses of SU are used. Although SU treatment offhand seems to constitute a logical choice of treatment in MODY, due to beta cell dysfunction, the risk of hypoglycaemia is a clinical drawback due to potential suboptimal glycaemic control and decreased patient compliance. In a recent study, in which patients with MODY3 were exposed to physical activity (light cycling for 30 minutes approximately 2 hours after meal ingestion), hypoglycaemia was observed in 40% of subjects treated with short-acting SU (glibenclamide) with one patient experiencing hypoglycaemia for 12 hours.

Glucagon-like peptide-1 (GLP-1) is an incretin hormone, which is secreted from endocrine L cells of the small intestine in response to nutrients in the gut lumen. GLP-1 conveys an insulinotropic effect through GLP-1 receptors (GLP-1R) on pancreatic beta cells thereby decreasing plasma glucose (PG). Moreover, GLP-1 inhibits the secretion of glucagon from pancreatic alpha cells, which further contributes to lowering of the PG levels. Both of these effects are strictly glucose-dependent (more pronounced at higher PG levels) and the effects cease as PG levels reaches values below 4-5 mM. Therefore, the hormones keep PG at normal levels without increasing the risk of hypoglycaemia. In addition, GLP-1 inhibits gastrointestinal motility including gastric emptying and leads to a centrally-mediated inhibition of appetite resulting in reduced food intake. Thus, GLP-1 is essential for glycaemic control. The GLP-1R agonist, liraglutide (Victoza®), has 97% homology to the naturally occurring GLP-1 hormone, but has a longer half-life (11-15 hours).

Since the effects of the incretin hormones are strictly glucose-dependent, treatment with GLP-1R agonists is rarely associated with hypoglycaemia. Thus, the current study aims to elucidate whether liraglutide (Victoza®) could be a safe and efficacious new treatment modality for patients with MODY.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian above 18 years of age
* Well characterised MODY3
* Body mass index (BMI) > 19 kg/m2
* Normal haemoglobin (males > 8.2 mM, females > 7.2 mM)
* Normal blood pressure (< 160/100 mmHg)
* Informed consent
* Capability to perform a light cycling test (heart rate 100-120 beats per minute during 30 minutes)
* Females: use of anticonception (IUC or hormonal)

Exclusion Criteria:

* Heart failure: New York Heart Association class III-IV
* Uraemia, end-stage renal disease, or any other cause of impaired renal function with s-creatinine > 130 µM and/or albuminuria
* Liver disease (alanine amino transferase (ALAT) and/or aspartate amino transferase (ASAT) > 2 × upper normal serum levels)
* Anaemia
* Acute or chronic pancreatitis
* Stroma or thyroid cancer
* Pregnancy or breast feeding
* Inability to complete the study
* Treatment naïve patients with HbA1c < 7.0 %
* Treatment with medicine that can not be paused for 12 hours
* Known allergic reaction to study medication
* Intention to become pregnant
* Unwillingness to complete the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Fasting Plasma Glucose | 14 weeks
  Glycaemic control will be evaluated by FPG monitored twice weekly, 7-point PG profiles every two weeks and 3 blinded 48-hour continuous PG profiles (before randomisation and at the end of both treatment periods). The patients who will be their own controls, will randomly be assigned (after one week washout of usual antidiabetic treatment) to receive either liraglutide or glimepiride for 6 weeks, and after another one-week washout period treated with the opposite treatment for 6 weeks.

SECONDARY OUTCOMES:
Serum Fructosamine | 14 weeks
  Fructosamine is a time-averaged indicator of PG levels. It reflects the total amount of glycated proteins such as glycohaemoglobin and glycoalbumin in a blood sample. The turnover of serum proteins (albumin has a half-life of 19 days) is less than that of haemoglobin, and therefore fructosamine determinations provide a means of monitoring patient blood glucose status over a shorter period (1-3 weeks) than glycohaemoglobin (6-8 weeks).
Hypoglycemic events | 14 weeks
  Hypoglycaemic events will be reported by the patient in a diary. During cycling tests patients will be tested further according to hypoglycaemia. Mild hypoglycaemia is defined as episodes with symptoms of hypoglycaemia familiar to the patient and managed solely by the patient. Events of severe hypoglycaemia are defined as episodes with symptoms of hypoglycaemia with need for assistance from another person.
Plasma concentrations of insulin and C-peptide | 14 weeks
  Postprandial responses of incretin hormones and beta cell function (assessed as fasting proinsulin-to-insulin ratio) will be evaluated during three standardised 4-hour meal tests (at baseline and in the end of each treatment period).
Plasma glucagon | 14 weeks
  Postprandial responses of incretin hormones and beta cell function (assessed as fasting proinsulin-to-insulin ratio) will be evaluated during three standardised 4-hour meal tests (at baseline and in the end of each treatment period).
Plasma concentrations of incretin hormones | 14 weeks
  Postprandial responses of incretin hormones and beta cell function (assessed as fasting proinsulin-to-insulin ratio) will be evaluated during three standardised 4-hour meal tests (at baseline and in the end of each treatment period).

CONTACTS AND LOCATIONS:
Overall Officials: Signe H Østoft, MD, Principal Investigator — Diabetes Research Division, University Hospital Gentofte, Denmark
Locations (1):
- Diabetes research Division, University Hospital Gentofte, Hellerup, Denmark

REFERENCES:
- [Derived] Ostoft SH, Bagger JI, Hansen T, Pedersen O, Faber J, Holst JJ, Knop FK, Vilsboll T. Glucose-lowering effects and low risk of hypoglycemia in patients with maturity-onset diabetes of the young when treated with a GLP-1 receptor agonist: a double-blind, randomized, crossover trial. Diabetes Care. 2014 Jul;37(7):1797-805. doi: 10.2337/dc13-3007. PMID 24929431